CLINICAL TRIAL: NCT05489601
Title: Prove the Feasibility of a Non-invasive Means to Identify Temporary Neurological Impairment Resulting From the Use of a Commonly Prescribed Opioid by Identifying an Oculomotor Biosignature Associated With Temporary Neurologic Impairment in Pain-free Opioid-naïve Subjects, and to Initiate the Development of Such a Signature.
Brief Title: Non-intrusive Detection of Temporary Neurologic Impairment by Opioids
Status: Completed | Type: Observational
Sponsor: Zxerex Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: OpioidsPhaseI
Record Dates: First submitted 2022-07-26; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Impairment by Opioids
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants: * Adults between 21 and 59 years of age.
  * Males and females; women must practice an effective form of birth control (condoms, diaphragm, birth control pill, IUD).
  * Subjects have taken an opioid prescription for pain management within the prior 24 months and have not used any opioids during the preceding 30 days.
  * Subjects are required to have a negative urine drug test. At any point during the study, If a subject is found to have a positive drug test, the subject will be discontinued from the study.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Oxycodone in 5mg increments up to a maximum of 10mg

SUMMARY:
The investigators aim to prove the feasibility of a non-invasive means to identify temporary neurological impairment resulting from the use of a commonly prescribed opioid by identifying an oculomotor biosignature associated with temporary neurologic impairment in pain-free opioid-naïve subjects, and to initiate the development of such a signature. The investigators also sought to establish the presence of a dose-dependent biosignature for opioid impairment.

DETAILED DESCRIPTION:
To determine the detrimental effects of opioid intoxication on normal oculomotor function, the investigators will collect data from up to 25 subjects before and during oxycodone induced intoxication. A within-subjects design will be used, and subjects will be tested under conditions of no dose (placebo), low dose, and high dose. Subjects will be tested during 3 sessions (baseline, placebo, oxycodone); separated by 7 days to allow for complete washout of any drug that was administered. Subjects will perform tests of visual fixation, saccade speed and saccade accuracy, cognitive control over saccades, cognitive control over visual scanning, and visual pursuit. Eye movement data will be collected using an SR Research EyeLink 1000 Plus eye tracking system.

Analysis of the data will be performed by comparing each subject state against the baseline measurements, where baseline represents an unimpaired subject state. Based on prior work with marijuana intoxication, the investigators expect that this data and analysis will successfully reveal a constellation of oculomotor dynamics that can be used to classify whether an individual is or is not currently impaired by oxycodone. Based on published studies, the investigators anticipate these changes will generalize across the opioid class, creating a biosignature of opioid impairment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 21 and 59 years of age.
* Males and females; women must practice an effective form of birth control (condoms, diaphragm, birth control pill, IUD).

Exclusion Criteria:

* Prior use of any opioids during the preceding 30 days.
* Positive urine drug test for any drug at any point during the study.
* Pregnancy

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants recruited from area local to Scottsdale, Arizona
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Eye movement velocity | 1 hour post-dose for 3 hours across 3 sessions, minimum 48 hours between sessions.
  Eye position over time is recorded and tracked using a specialized eye-tracking camera system during a battery of visual tests under control and oxycodone challenge conditions. This data is converted to a velocity measure as millimeters per second (mm/second) and then converted to an angular velocity as degrees of visual angle per second (dva/second).
Pupil area change | 1 hour post-dose for 3 hours across 3 sessions, minimum 48 hours between sessions.
  Changes in pupil area are recorded over time using specialized a eye-tracking camera system.
  Screen illumination is abruptly changed from dark to maximum brightness and back while the pupils size is measured. The pupil area is represented in the units millimeters squared (mm^2).

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT05489601/Prot_SAP_000.pdf